CLINICAL TRIAL: NCT03780036
Title: A Randomised, Single Blind Study Assessing Radiological Outcomes for Massive Segmental Femoral Replacements Using Either Porous Collar or Porous Collar With HA
Brief Title: Megaprosthetic Implants the Next Generation (MING)
Acronym: MING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Adler Ortho, iEthos Medical Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0619-18-TLV
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Bone Neoplasm of Hip (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Random assignment of patients into one of the two study arms: porous collar magaprostheses or porous collar with HA megaprostheses.
Who Masked: Participant
Masking Description: The participant will not know which implant was used for segmental replacement of his or hear femur.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- porous collar (Experimental): Patients with neoplasm of femur bone who require segmental bone resection and replasement with a large prosthesis would receive an implant which collar (a circular part that comes into direct contact with the remaining bone) will be porous, to allow for bone ingrowth and stabilization of the implant.
  Interventions: Device: Megaprosthetic Implants the Next Generation (MING)
- porous collar with hydroxyapathite (Experimental): Patients with neoplasm of femur bone who require segmental bone resection and replasement with a large prosthesis would receive an implant which collar (a circular part that comes into direct contact with the remaining bone) will be porous and covered with hydroxyapathite particles, to allow for bone ingrowth and stabilization of the implant.
  Interventions: Device: Megaprosthetic Implants the Next Generation (MING)

INTERVENTIONS:
Device: Megaprosthetic Implants the Next Generation (MING) — Use of either porous of porous+hydroxyapathite collars.
  Other Names: Segmental bone replacement

SUMMARY:
This is an interventional randomized controlled trial that will compare patients who underwent segmental hip replacement using mega-implants with either porous collar or porous collar with HA. Patient recruitment will continue for 18 months. Parameters to be investigated are radiographic measures of bone incorporation into the implants, as well as patient functional outcomes. Clinical follow-up will last for 24 months for each patient.

DETAILED DESCRIPTION:
BACKGROUND The current surgical treatment of bone cancer patients requires usage of massive endoprosthetic bone implants. The incidence of aseptic loosening is a major cause of prosthesis failure in these patients. Exploring ways to reduce such failures would allow extending longevity of massive implants in a relatively young population.

Current published literature stipulates that osteointegration could improve longevity of massive implants. Evidence suggests that usage of osteointegrated hydroxyapatite (HA) coated collar would reduce the incidence of aseptic loosening around the cemented intramedullary stem in distal femoral bone prosthesis.

Our study aims to compare radiological outcome in 2 groups:

* A porous collar for either distal or proximal femoral replacements
* A porous collar with hydroxyapatite (HA) for either distal or proximal femoral replacements The porous collar will be manufactured by Adler Ortho using additive layer manufacturing technology.

STUDY OBJECTIVES The study will review the use of massive segmental replacements in the femur, which have a porous collar with and without HA.

Primary objectives:

The primary objective of the study will be to assess radiological outcome by assessing bony growth into the collar.

Secondary objectives The secondary objective will focus on assessing patient reported outcome measures (VAS pain score and other PROMS)

STUDY DESIGN

Patients will be identified in the outpatient setting as suitable for entry into the trial based on the inclusion and exclusion criteria as set out below.

Patients will be randomised into one of the two groups of the study, due to the nature of intervention this will be a single blind study.

Patients will undergo plain radiographs immediately post-operatively, at 6 months post-operatively, 12 months post-operatively and 24 months post-operatively. Standard protocol radiographs of the relevant limb will be taken in the antero-posterior (AP) and medial-lateral (ML) planes (x2 AP and x2 laterals to cover the prosthesis).

At 12 months and 24 months post-operatively patients will receive a CT scan (cover whole prosthesis, extended CT - knee, pelvis), which will be used to image bone growth within the porous collars.

For plain radiographs a scoring system for extra-cortical bone formation will be made according to Coathup et al, 2013. This will be quantified radiologically in four zones (medial and lateral aspects on AP radiographs; anterior and posterior aspects on ML radiographs). Extracortical bone separated from the implant by a clear radiolucent line is not considered in grown and will be scored 0. A score of 1 will represent extracortical bone (>5mm think and >1mm long) in contact with the implant surface in any of the four previously described zones. The maximum score will be 4, denoting extracortical bone growth in all four zones.

Patients identified and consented in clinic for entry into study. Randomisation prior to surgical date. Baseline X-ray and CT done pre-operatively as per current pre-operative guidelines.

Pre-operative bloods and joint aspiration done to definitively rule out infection in revision patients Pre-operative VAS pain score on admission

Joint replacement done - clarify antibiotic prophylaxis with surgeons - induction + extended post-operative antibiotic prophylaxis

Post-operative Toronto Extremity Salvage Score (TESS) to assess physical functioning for all patients. TESS repeated at 6, 12 and 24 months to assess progress post-operatively - correlating with radiographical findings.

Surgery related data including theatre time, intra-operative blood loss and intra- and post-operative complications will be recorded for all patients.

Immediate post-operative, 6, 12 and 24 monthly X-rays (x2 AP and x2 laterals to cover the prosthesis); 12 and 24 monthly CT (cover whole prosthesis, extended CT - knee, pelvis) X-rays and CT reported by scores calculated as previously described.

ELIGIBILITY:
Inclusion Criteria:

* Bone cancer patients requiring primary or revision femoral segmental replacements (excluding infections) and non-cancer patients requiring revision femoral segment replacement for aseptic loosening (excluding infections)
* Male or female, aged 18-80 years
* Participants willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Participants unwilling or unable to give informed consent for participation in the study
* Patients undergoing revision due to infection, identified by positive growth from joint aspiration OR elevated pre-operative inflammatory markers OR radiographical evidence of prosthetic joint infection
* Bone cancer patients presenting with pathological fractures requiring segmental femoral replacement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Bone incorporation | 24 months
  Radiographic evidence of bony growth into the collar

SECONDARY OUTCOMES:
Functional outcome - Visual Analogue Pain Scale | 24 months
  Reporting of pain levels (from 1 to 10)
Functional outcome - a physical functioning score | 24 months
  Toronto Extremity Salvage Score (TESS) for lower extremity

IPD SHARING:
Plan to Share IPD: No
De-identified data will be analyzed, and its summary will be shared with other researchers.

REFERENCES:
- [Background] Coathup MJ, Sanghrajka A, Aston WJ, Gikas PD, Pollock RC, Cannon SR, Skinner JA, Briggs TW, Blunn GW. Hydroxyapatite-coated collars reduce radiolucent line progression in cemented distal femoral bone tumor implants. Clin Orthop Relat Res. 2015 Apr;473(4):1505-14. doi: 10.1007/s11999-014-4116-6. Epub 2015 Jan 30. PMID 25634027
- [Background] Coathup MJ, Batta V, Pollock RC, Aston WJ, Cannon SR, Skinner JA, Briggs TW, Unwin PS, Blunn GW. Long-term survival of cemented distal femoral endoprostheses with a hydroxyapatite-coated collar: a histological study and a radiographic follow-up. J Bone Joint Surg Am. 2013 Sep 4;95(17):1569-75. doi: 10.2106/JBJS.L.00362. PMID 24005197
- [Background] Mumith A, Coathup M, Chimutengwende-Gordon M, Aston W, Briggs T, Blunn G. Augmenting the osseointegration of endoprostheses using laser-sintered porous collars: an in vivo study. Bone Joint J. 2017 Feb;99-B(2):276-282. doi: 10.1302/0301-620X.99B2.BJJ-2016-0584.R1. PMID 28148673